CLINICAL TRIAL: NCT01080573
Title: A Questionnaire Based Survey to Identify Issues With Patient Compliance and to Develop Solutions to Improve Rebif Compliance and Improve Patient Outcomes
Brief Title: Rebif Compliance Support Program - Assessing Needs in Multiple Sclerosis
Acronym: AIMS
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Dr Gillian Shepherd, Medical Director, Merck Serono Ltd. UK, an affiliate of Merck KGaA, Darmstadt, Germany
Other Study IDs: MMFM 100
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Rebif; Interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This 1-arm, open-label, multicentric, observational study aims to collect subject centric information in line with routine care. Subjects' expectations of therapy, side effect management and lifestyle may influence adherence to therapy. This survey aims to determine whether such factors and/or others affect the successful initiation and maintenance of Rebif therapy.

The data collected during this study will include information on the subject's treatment including expectations, experience, training and support. The results of the study will be used to understand the impact on subjects' compliance and tailor training and support services to subject's need. It will also be made available to other healthcare organisations involved in the subjects treatment.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating disease of the central nervous system and is one of the most common causes of neurological disability in young adults. It is characterised by multifocal, recurrent attacks of neurological symptoms and signs with variable recovery. Eventually the majority of subjects develop a progressive clinical course. It is important to carefully initiate and maintain subjects with MS on therapy. Information will be gathered in a structured way which will enable easier identification of any subgroups of subjects who may be at risk of poor compliance. These risk groups could possibly include groups with particular attributes such as poor information at the start of treatment, unrealistic expectations or a particular life style. This study will be conducted during the contact with the subject necessary to deliver the homecare service. Participants will be contacted by Bupa Home Healthcare Multiple Sclerosis subject coordinators by telephone to conduct specific questionnaires during the 4 stages of the subject's treatment i.e. pre-installation of treatment, post installation of treatment, monthly pre delivery of drug and at a subject's end treatment.

OBJECTIVES

* To collect subject centric information in line with routine care including subject's expectations of therapy, side effect management and lifestyle may influence adherence to therapy
* To determine whether such factors and/or others affect the successful initiation and maintenance of Rebif therapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been prescribed Rebif and referred to Bupa Home Healthcare service by one of the participating referring centres

Exclusion Criteria:

* Subject unwilling to give informed consent
* Subjects visiting private clinics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have been prescribed Rebif and referred to Bupa Home Healthcare service by one of the participating referring centres.
Sampling Method: Non-Probability Sample
Enrollment: 1257 (Actual)
Dates: Start 2007-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Discontinuation of Rebif treatment (yes or no) | Data collection is expected to end 3 months after last subject is recruited

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gillian Shepherd, MD MRCP, Study Director — Merck Serono UK Ltd
Locations (1):
- Bupa Home Healthcare, Harlow, Essex, United Kingdom